CLINICAL TRIAL: NCT02057146
Title: Endoscopic Evaluation of Premalignant Lesions in the Biliary Tract and Pancreatic Ducts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1658-31; 2013/1658-31 (Other: Ethical Review Board)
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Benign Neoplasm of Liver and/or Biliary Ducts; Neoplasm of Uncertain Behavior of Biliary System; Benign Neoplasms of the Pancreas; Neoplasms of the Pancreas
Keywords: PSC; mother-baby endoscopy; ERCP; IPMN
MeSH Terms: interventions — Duodenoscopy; Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mother-baby endoscopy (Experimental): Spyglass mother-baby endoscopy in conjunction with ERCP
  Interventions: Procedure: Duodenoscopy, pancreatoscopy, cholangioscopy, confocal microscopy

INTERVENTIONS:
Procedure: Duodenoscopy, pancreatoscopy, cholangioscopy, confocal microscopy — The intervention consists of mother-baby endoscopy of the bile and/or pancreatic duct with visual inspection, confocal laser microscopy, collection of fluid for cytology, and eventually biopsy.
  Other Names: Spyglass; Cellvizio; pCLE

SUMMARY:
Single operater pancreatico-cholangioscopy is performed through the working channel of conventional duodenoscopes. A visual evaluation of the biliary and pancreatic ductal systems is completed and obvious or suspicious macroscopic lesions are targeted by biopsy forceps.

Evaluation of the usefulness of probe based confocal laser endomicroscopy in the evaluation of suspected premalignant lesions in the biliary duct and in the pancreas.

DETAILED DESCRIPTION:
Diagnosis of early preneoplastic lesions is always a problem, but especially when it comes to hidden organs such as the bile ducts and the pancreas. The recent developments in endoscopy encompass mini endoscopes (mother-baby; "Spyglas®"), which allow visualization of the bile ducts and the pancreas and the possibility to take biopsies under direct vision. An even newer technique is an adaptation of the existing confocal laser scanning microscopy (CLSM) to a small probe, which fits into the 1 mm working channel of the Spyglas. This application of CLSM was coined probe-based confocal laser endomicroscopy (pCLE).

It is the aim of this project to systematically and prospectively evaluate the usefulness of pCLE in two distinct patient groups: patients with PSC prone to develop a bile duct cancer (CCC) and patients with chronic pancreatitis/family history of pancreatic cancer prone to develop pancreatic cancer or have suspected IPMN.

Patients&Methods Patients with suspected diagnosis of PSC who have to undergo ERCP for diagnosis or therapy or suspected CCC will receive Spyglass investigations under a current clinical protocol. The investigators will add pCLE to these patients.

Patients with chronic (hereditary) pancreatitis and suspected malignancy, patients with suspected premalignant lesions (e.g. IPMN), and individuals at risk from familiar pancreatic cancer syndromes who under the surveillance (MRCP with secretin) demonstrate a pancreatic pathology will undergo ERCP with Spyglass as a diagnostic procedure. In these patients, the investigators will add pCLE.

Spyglass will be introduced during ERCP and the ducts will be visually inspected. In areas of stenosis and/or suspected pathology, pCLE will be executed. Finally, these areas will be biopsied, if possible. Bile and pancreatic juice will be taken for cytology and molecular analysis. Diagnostic yield and accuracy will be determined of ERCP (x-ray), Spyglas, CLSM, and histology (PAD).

This will be firstly an explorative study because the diagnostic criteria for assessing malignancy with CLSM are under development and the investigators group as one of the few doing Spyglas routinely will contribute to establishing such criteria. For statistical calculations, a total of 100 patients will be necessary. It is their plans to do this prospectively together with several centers once the diagnostic criteria are set in order to fulfill the statistical needed numbers.

Significance An early diagnosis of both CCC developing in PSC patients and PDAC developing in CP, IPMN patients or individuals with familiar history of PDAC would allow us to treat these patients in good time with surgery or transplantation (LTX). This, in turn, is the only way to improve the diagnosis of these tumors as the have amongst the worst prognosis of all solid tumors in man.

ELIGIBILITY:
Inclusion Criteria:

* Suspicious lesions of the hepatobiliary pancreatic duct systems.

Exclusion Criteria:

* Unwillingness to participate
* Unfit for the investigation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Accuracy of single operator endoscopy plus pCLE in the biliary and pancreatic ductal system diagnosing premalignant and malignant lesions. | Two years
  Beside the safety, technical feasibility and efficacy, we will record and calculate the diagnostic accuray by comparing the outcome of Spyglass/pCLE (endoscopic judgement) with histology (biopsy) and eventual surgical pathology.
  Outcome measures will be 1) diagnosis of malignant/suspicious lesion by Spyglass and/or pCLE versus final diagnosis with biopsy (Spyglass, other) and/or surgical pathology (resection).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Löhr, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Arnelo U, Albiin N, Enochsson L, Meisner S, Permert J, Lundell L. Endoscopic evaluation of the pancreatic duct system: opportunities offered by novel technology. Scand J Gastroenterol. 2007 Aug;42(8):1018-20. doi: 10.1080/00365520601101526. PMID 17613934
- [Result] Arnelo U, Valente R, Scandavini CM, Halimi A, Mucelli RMP, Rangelova E, Svensson J, Schulick RD, Torphy RJ, Fagerstrom N, Moro CF, Vujasinovic M, Matthias Lohr J, Del Chiaro M. Intraoperative pancreatoscopy can improve the detection of skip lesions during surgery for intraductal papillary mucinous neoplasia: A pilot study. Pancreatology. 2023 Sep;23(6):704-711. doi: 10.1016/j.pan.2023.06.006. Epub 2023 Jun 12. PMID 37336668
- [Result] Lohr JM, Lonnebro R, Stigliano S, Haas SL, Swahn F, Enochsson L, Noel R, Segersvard R, Del Chiaro M, Verbeke CS, Arnelo U. Outcome of probe-based confocal laser endomicroscopy (pCLE) during endoscopic retrograde cholangiopancreatography: A single-center prospective study in 45 patients. United European Gastroenterol J. 2015 Dec;3(6):551-60. doi: 10.1177/2050640615579806. PMID 26668748